CLINICAL TRIAL: NCT05704712
Title: Empirical Testing of a Widely Available Insurance-based Monetary Incentive Program for Exercise: A Randomized Trial
Brief Title: Exercise Incentives for YMCA Based Exercise
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, David M. Williams, Professor, Brown University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: R01CA262894 (NIH); R01CA262894 (NIH)
Record Dates: First submitted 2023-01-09; First posted 2023-01-30 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Physical Inactivity
Keywords: Incentives; Motivation
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Message 1 - $100 (Experimental): Participants are offered an incentive of $100 to complete 50 exercise sessions at the YMCA within 6 months (Description of incentive 1)
  Interventions: Behavioral: Monetary Incentives
- Message 2 - $100 (Experimental): Participants are offered an incentive of $100 to complete 50 exercise sessions at the YMCA within 6 months (Description of incentive 2).
  Interventions: Behavioral: Monetary Incentives
- Message 1 - $200 (Experimental): Participants are offered an incentive of $200 to complete 50 exercise sessions at the YMCA within 6 months (Description of incentive 1).
  Interventions: Behavioral: Monetary Incentives
- Message 2 - $200 (Experimental): Participants are offered an incentive of $200 to complete 50 exercise sessions at the YMCA within 6 months (Description of incentive 2).
  Interventions: Behavioral: Monetary Incentives
- Control (No Intervention): Participants complete all assessments, and are eligible to receive compensation for participating in the research components of the study.

INTERVENTIONS:
Behavioral: Monetary Incentives — Monetary incentives, provided in the form of pre-loaded Visa debit cards are provided to encourage exercise.
  Arms: Message 1 - $100; Message 1 - $200; Message 2 - $100; Message 2 - $200

SUMMARY:
The investigators will conduct a randomized controlled trial to test financial incentive programs (versus control) to promote physical activity among 330 adults who have a YMCA membership. Participants will have the opportunity to earn up to $100 or $200 (depending on the condition they are assigned to) for attending at least 50 sessions at the YMCA over 6 months. Participants will have two 6-month windows during which they will have the opportunity to earn the incentive. In addition to the incentives, participants will complete research assessments every 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. A current member, or willing to become a current member of one of the following branches of the YMCA:

   1. Bayside Family YMCA (Barrington, RI)
   2. Cranston YMCA (Cranston, RI)
   3. East Side/Mt. Hope YMCA (Providence, RI)
   4. Kent County YMCA (Warwick, RI)
   5. Newman YMCA (Seekonk, MA)
   6. South County YMCA (South Kingston, RI)
2. Age 18 years or older
3. Physically capable of engaging in exercise

Exclusion Criteria:

1. Not a current member, and unwilling to become a member of one of the above listed YMCA branches.
2. Under age 18.
3. Physically incapable of exercise
4. Doctor has recommended that you should not exercise because of a current health condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2023-03-16 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Number of YMCA visits | Baseline, 6 months, 12 months, 24 months
  Number of sessions (max 1 per day) a person signs into the YMCA

SECONDARY OUTCOMES:
Change in Accelerometry | Measured at baseline, and months 3, 6, 9, and 12.
  Minutes of physical activity weighted by intensity, expressed in metabolic equivalent (MET) minutes per week as determined by accelerometers (Actigraph [model wGT3x-BT]) worn during one-week periods.
Change in Self-report physical activity (Godin) | Measured at baseline, and months 3, 6, 9, and 12.
  Self-reported minutes of leisure time physical activity (inside and outside the YMCA) per week weighted by intensity

OTHER OUTCOMES:
Change in Self-Reported Habit of Physical Activity Questionnaire | Measured at baseline, and months 3, 6, 9, and 12.
  Measures a person's habits regarding exercise, with a minimum value of 1 and a maximum value of 7, higher scores indicate a stronger habit.
Change in Anticipated Regret Questionnaire | Measured at baseline, and months 3, 6, 9, and 12.
  Measures a person's anticipated feelings of remorse if they do not do exercise, or achieve the incentives, on a scale from 1-11, with higher scores indicating more anticipated regret.
Change in Opportunity Questionnaire | Measured at baseline, and months 3, 6, 9, and 12.
  Measures a person's opportunity to do regular aerobic physical activity, with scores ranging from 1-7, and higher scores indicating more opportunity for physical activity.
Change in Capability Questionnaire | Measured at baseline, and months 3, 6, 9, and 12.
  Measures a person's physical and psychological capability to do regular aerobic physical activity with scores ranging from 1-7, and higher scores indicating more capability for physical activity.
Change in Exercise Facility Use Questionnaire | Measured at baseline, and months 3, 6, 9, and 12.
  Measures access and membership to fitness facilities.
Change in Physical Activity Hedonic/Reflective Motivation | Measured at baseline, and months 3, 6, 9, and 12.
  Measures the extent to which a person's motivation for physical activity is rooted in reflective and/or hedonic processes. There are two subscales. The hedonic subscale ranges from 0-10, with higher scores indicating more hedonic motivation for physical activity. The reflective subscale ranges from 0-10 with higher scores indicating more reflective motivation for physical activity.
Change in Subjective Social Status | Measured at baseline, and months 3, 6, 9, and 12.
  Measures a person's perception of their subjective social status
Change in Reward Responsiveness | Measured at baseline, and months 3, 6, 9, and 12.
  Measures the extent to which a person is responsive to external rewards
Change in Consideration of Future Consequences | Measured at baseline, and months 3, 6, 9, and 12.
  Measures the extent to which a person considers the future (delayed) consequences of their actions
Change in Delay Discounting | Measured at baseline, and months 3, 6, 9, and 12.
  Measures the extent to which a person discounts future rewards and prioritizes immediate rewards
Change in Loss Aversion | Measured at baseline, and months 3, 6, 9, and 12.
  Measures the extent to which a person chooses actions in an attempt to avoid experiencing losses
Change in Overall Health (SF-12 Survey) | Measured at baseline, and months 3, 6, 9, and 12.
  Measures a person's perception of their overall health and quality of life, scores range from 1-5 with higher scores indicating poorer health outcomes.
Change in Quality of Life and Health Status (EQ-5D-5L) | Measured at baseline, and months 3, 6, 9, and 12.
  The EQ-5D-5L comprises a short descriptive system questionnaire and a visual analogue scale (EQ VAS) that are cognitively undemanding, taking only a few minutes to complete. The questionnaire provides a simple descriptive profile of a respondent's health state. The EQ VAS provides an alternative way to elicit an individual's rating of their own overall current health. When the descriptive system profile is linked to a 'value set', a single summary index value for health status is derived that can be used in economic evaluations of health-care interventions. A value set provides values (weights) for each health state description according to the preferences of the general population of a country/region. Value sets for the EQ-5D-5L and 3L versions are available in a large and growing number of countries.
Change in Absenteeism and Presenteeism | Measured at baseline, and months 3, 6, 9, and 12.
  Measures the amount of time a person worked and was expected to work in the past 7-28 days; and their perceived job performance when at work

CONTACTS AND LOCATIONS:
Overall Officials: David M Williams, Ph.D., Principal Investigator — Brown University School of Public Health; Omar Galarraga, Ph.D., Principal Investigator — Brown University School of Public Health
Locations (1):
- Brown University, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared with interested parties after all of the initial study analyses and outcomes have been published.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available 1 year after study completion.
Access Criteria: All data access requests will be reviewed by a panel prior to acceptance

REFERENCES:
- [Derived] Williams DM, Bohlen LC, Dunsiger S, Ayala-Heredia V, Griffin E, Dionne L, Wilson-Barthes M, Unick J, LaRowe LR, Galarraga O. Testing an insurance-based monetary incentive program for exercise: RCT design and rationale. Contemp Clin Trials. 2023 Dec;135:107382. doi: 10.1016/j.cct.2023.107382. Epub 2023 Nov 5. PMID 37935304

DOCUMENTS (1):
  • Informed Consent Form (2022-12-12): https://cdn.clinicaltrials.gov/large-docs/12/NCT05704712/ICF_000.pdf